CLINICAL TRIAL: NCT05826600
Title: A Phase I/Ib Dose Escalation and Cohort Expansion Study of OMX-0407 a Salt-inducible Kinase Inhibitor in Patients With Previously Treated Unresectable Solid Tumours
Brief Title: A Study of OMX-0407 in Patients With Previously Treated Solid Tumours That Can't be Removed Surgically
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: iOmx Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: OMX-0407-101
Record Dates: First submitted 2023-03-14; First posted 2023-04-24 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor
Keywords: Renal Cell Carcinoma; Angiosarcoma
MeSH Terms: conditions — Carcinoma, Renal Cell; Hemangiosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OMX-0407 - Escalation Phase (Experimental): A starting daily dose of 20 mg OMX-0407 per participant split into twice daily 10 mg.
  Dose escalation will be determined by the safety monitoring committee. Dose for expansion will be determined by the safety monitoring committee.
  Interventions: Drug: OMX-0407
- OMX-0407 - Expansion Phase (Phase Ib) (Experimental): A dose of 100 mg OMX-0407 will be orally administered twice daily.
  Interventions: Drug: OMX-0407

INTERVENTIONS:
Drug: OMX-0407 — Dose escalation, Dose expansion

SUMMARY:
The main purpose of the dose escalation phase of the study is to determine the safety of different doses of OMX-0407.

The dose expansion (phase Ib) part of the study will evaluate efficacy, safety and tolerability at a dose determined in the dose escalation,

ELIGIBILITY:
General Inclusion Criteria for Cohort Expansion Phases

1. Age ≥18 years (≥16 years for the AS expansion cohort) and willing to provide informed consent for the study.
2. Cytological or pathological confirmation of advanced cancer.
3. Subjects treated in three subject cohorts onwards will be required to provide either archival tumour material or be willing to undergo a core biopsy to provide tumour material during screening.
4. Subjects should have completed or be unsuitable for licensed therapies for their primary cancer unless such therapies are not available according to local practice - for example not reimbursed or included in treatment guidelines. All subjects must have received at least one previous line of systemic therapy for the tumour type under investigation. Subjects who have declined treatment or according to their treating physician are unsuitable for an existing licensed therapy are eligible for the study.
5. Eastern Cooperative Oncology Group (ECOG) Performance status 0, 1 or 2. Subjects treated in the cohort expansion phase of the study should have an ECOG Performance status of 0 or 1.
6. Able to swallow oral medication with no existing evidence of underlying gastrointestinal malabsorption or abnormal gastrointestinal transit.
7. For female subjects and male partners of childbearing potential, willingness and able to use two forms of highly effective contraception methods (e.g., oral contraceptive and condom, intra-uterine device, and condom) while on study and for 30 days after the last study treatment. For male subjects and female partners of childbearing potential, willingness and able to use two forms of highly effective contraception methods (e.g., oral contraceptive and condom, intra-uterine device, and condom) while on study and for 3 months after the last study treatment. Women who last experienced menses more than one year previously or who have undergone bilateral ovariectomy, hysterectomy or tubal ligation which is documented in their medical notes do not require to use contraception during or after treatment with OMX-0407. Male subjects who have previously undergone vasectomy are not required to use contraception.
8. All toxicity from previous anti-cancer therapy including radiotherapy must have recovered to either Grade I or stable Grade II (CTCAE v5).
9. Subjects should have at least evaluable tumour by Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 criteria. Subjects treated in the Cohort Expansion phases of the study should have measurable disease.

Additional Inclusion Criteria For Cohort Expansion Phase: ccRCC

1. Prior histological confirmation of clear cell renal cell carcinoma. In the case of mixed histology in order to be eligible at least 70% of reviewed tumour should be of clear cell histology.
2. Subjects with known renal vascular involvement should be on stable anticoagulation at the start of treatment with OMX-0407. Tumour/skin biopsies should be performed prior to the onset of anticoagulation.
3. Previous treatment must include PD-1 blockade and VEGFR inhibition.

Additional Inclusion Criteria for Cohort Expansion Phase: AS

1. Clinical and histopathological confirmation of advanced/metastatic or unresectable visceral AS, cutaneous AS secondary to radiotherapy or other cutaneous AS.
2. Subjects should have progressive disease
3. Subject has received at least one prior line of systemic therapy for metastatic or unresectable disease which must have included a taxane or an anthracycline.
4. Willingness to undergo serial tumour biopsies before and during study treatment.

Patient will still be eligible if the investigator deems the biopsy procedure to be an unacceptable health risk to the patient.

General Exclusion Criteria for Cohort Expansion Phases

1. Untreated CNS metastases. Subjects with CNS metastases that have completed treatment at least two weeks previously and have either an unchanging or no neurological deficit whilst not receiving corticosteroid therapy are eligible. Subjects with known CNS metastases must have received CNS directed therapy and not systemic therapy alone to be eligible for the study.
2. Either Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) > 2.5 upper limit of normal (ULN) unless in the presence of hepatic metastases when AST or ALT as high as 5 ULN is acceptable. Serum bilirubin > 1.5 ULN unless in the presence of hepatic metastases when serum bilirubin as high as 3 x ULN is acceptable. Subjects with isolated increases in alkaline phosphatase (ALK) are eligible for the study.
3. Prothrombin Time or equivalent such as international normalized ratio (INR) or the Quick test > 1.5 ULN.
4. Activated Partial Thromboplastin Time (PTT) > 1.5 ULN.
5. Chronic anticoagulant therapy that cannot be discontinued for tumour biopsy if necessary.
6. Previous biological or unlicensed anticancer therapy within five half-lives or thirty days of treatment - whichever is shortest.
7. Prior cytotoxic chemotherapy in the preceding three weeks.
8. Persistent fever or other signs of uncontrolled infection.
9. Creatinine clearance by Cockcroft-Gault formula or local equivalent < 30 ml/min.
10. Allergy to OMX-0407 or any of its excipients.
11. Personal or family history of long QT syndrome or sudden death.
12. Family or personal history of ventricular arrythmia. Known untreated aberrant preexcitation pathways such as Wolf-Parkinson-White syndrome. Ongoing atrial fibrillation unless the ventricular rate is controlled by medical therapy.
13. Unstable hypertension requiring changes in antihypertensive medication within the preceding three months, Myocardial Infarction or Cerebrovascular accident within the preceding three months. Cardiac failure New York Heart Association (NYHA) Grade III or IV.
14. Abnormal echocardiogram (ECHO) according to investigational site criteria including a normal Ejection Fraction.
15. QTc interval after Fridericia correction of greater than 450 ms (man) or 460 ms (woman) (mean of three readings performed at least five minutes apart).
16. Second degree Atrioventricular block or cardiac pacemaker.
17. Subject must have fully recovered from major surgery such as thoracotomy. Open biopsy or insertion of a venous access device does not constitute major surgery.
18. Known active Hepatitis B (HBV) or C (HCV) including subjects receiving antiviral therapy. Subjects with a history of hepatitis are eligible for the study if they are positive for anti-HBs or do not have detectable HCV mRNA at least six weeks from completing antiviral therapy.
19. Ongoing disabling systemic disease such chronic obstructive pulmonary disease (COPD) or depression or other psychiatric illnesses which may reduce study compliance.
20. Ongoing drug dependence or parenteral substance abuse.
21. Concurrent use of medications at risk of Torsade de pointes under normal clinical usage.
22. Live vaccinations in the preceding four weeks.
23. Subjects who have received treatment for another malignancy in the preceding three years other than squamous cell or basal cell carcinoma of the skin, Carcinoma In Situ of the uterine cervix, Ductal Carcinoma In Situ of the breast, non-muscle invasive carcinoma of the bladder, melanoma in situ or adenocarcinoma of the prostate (Gleason score of five or less).
24. Myelosuppression defined as any of the below:

    Haemoglobin <9.5 g/dl White Cell Count <2 x 1000 per μl Neutrophils <1.5 x 1000 per μl Platelets <75 000 per μl Independent of haematopoietic growth factors and transfusion
25. Receipt of any other investigational anticancer agent within 28 days prior to first administration of OMX-0407.
26. Female subjects must not be pregnant or breast feeding.

Additional Exclusion Criteria for Cohort Expansion Phase: ccRCC 1. Uncontrolled hypertension defined as persistent BP greater than Diastolic 90 mm Hg and Systolic 150 mm Hg

Additional Exclusion Criteria for Cohort Expansion Phase: ccRCC and AS

1. More than 3 previous lines of therapy in an unresectable or metastatic setting.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Identify Dose Limiting Toxicities | 4 weeks (1 cycle)
  Incidence of dose limiting toxicities at each dose level
Identify objective response rate | Every 12 weeks (3 cycles)
  Number of objective responses of OMX-0407 in patients with Renal Cell cancer, Non small cell lung cancer, urothelial cancer and angiosarcoma

SECONDARY OUTCOMES:
Maximum Tolerated Dose | evaluated up to approximately 3 years
  Identify the maximum tolerated dose and recommended dose for Phase II based on toxicities at each dose level
Investigate the safety and tolerability of OMX-0407 | through study completion, estimated up to approximately 3 years
  Incidence and severity of adverse events at each dose level
Pharmacokinetics (Cmax) of OMX-0407 | evaluated up to approximately 3 years
  Maximum observed plasma concentration
Pharmacokinetics (Tmax) of OMX-0407 | evaluated up to approximately 3 years
  Time of maximum observed plasma concentration
Pharmacokinetics (AUClast) of OMX-0407 | evaluated up to approximately 3 years
  Area under the plasma concentration-time curve from time of dosing to the last quantifiable timepoint
Pharmacokinetics (AUCinf) of OMX-0407 | evaluated up to approximately 3 years
  Area under the plasma concentration-time curve from time of dosing to infinity
Pharmacokinetics (% extrapolated-AUCinf) of OMX-0407 | evaluated up to approximately 3 years
  The percentage of AUCinf derived via extrapolation from Tlast
Pharmacokinetics (t½) of OMX-0407 | evaluated up to approximately 3 years
  Terminal elimination half-life
Measure Duration of Response | every 12 weeks (3 cycles)
  Determine the median duration of response according to RECIST 1.1
Measure Progression Free Survivial | every 12 weeks (3 cycles)
  Determine the median time for progression free survival
Measure Overall Response Rates | every 12 weeks (3 cycles)
  Determine the overall number of responses
Measure Overall Survival | every 12 weeks (3 cycles)
  Determine the survival times of patients
Assess Quality of Life | Every 4 weeks (1 cycle)
  Determine changes in quality of life

OTHER OUTCOMES:
Explore Target Kinase Inhibition | evaluated up to approximately 3 years
  Changes in selected kinase activity and T cell subset analysis in circulating peripheral blood cells, skin and tumour biopsy material
Explore and characterize the metabolites of OMX-0407 | evaluated up to approximately 3 years
  Analysis of metabolites presence in serum blood samples
Explore associations of pre-treatment tumour biology with treatment outcome | evaluated up to approximately 3 years
  Analyse the molecular features pre and post treatment

CONTACTS AND LOCATIONS:
Locations (24):
- Belgium (4):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - CHU de Liège, Liège
  - ZAS Augustinus Afdeling Oncologische Research, Wilrijk
- France (8):
  - UNICANCER-Institut Bergonie - Nouvelle-Aquitaine, Bordeaux
  - Universite de Lyon - Centre Leon-Berard (CLB), Lyon
  - Assistance Publique Hopitaux de Marseille- Hopital de La Timone, Marseille
  - Institut du Cancer Montpellier (ICM), Montpellier
  - Institut de Cancerologie de Ouest (ICO) - Saint-Herblain, Nantes
  - UNICANCER - Centre Oscar Lambret, Nantes
  - Gustave Roussy - Institut Gustave Roussy, Paris
  - CHU de Toulouse, Toulouse
- Spain (12):
  - ICO Hospitalet, L'Hospitalet de Llobregat, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitario Vall d'Hebrón, Barcelona
  - NEXT Oncology - Hospital Quironsalud Barcelona, Barcelona
  - Hospital Universitario Gregorio Marañon, Madrid
  - Clínica Universidad de Navarra, Madrid
  - MD Anderson Cancer Center, Madrid
  - START Madrid - Hospital Fundacion Jimenez Diaz, Madrid
  - Centro Integral Oncológico Clara Campal, Madrid
  - NEXT Oncology - Hospital Universitario Quironsalud, Madrid
  - Clínica Universidad de Navarra, Pamplona
  - Hospital La Fe de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR